CLINICAL TRIAL: NCT00414401
Title: Clinical Reminders in Test Reports to Improve Guideline Compliance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: IIR 01-108
Record Dates: First submitted 2006-12-19; First posted 2006-12-21 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2006-12

CONDITIONS: Heart Failure, Congestive
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other)
  Interventions: Behavioral: Clinical Reminder

INTERVENTIONS:
Behavioral: Clinical Reminder

SUMMARY:
Although beta-blockers are known to prolong survival for patients with reduced left ventricular ejection fraction, their use in the community and the VA is suboptimal.

DETAILED DESCRIPTION:
Background:

Although beta-blockers are known to prolong survival for patients with reduced left ventricular ejection fraction, their use in the community and the VA is suboptimal.

Objectives:

To determine if a reminder attached to the echocardiography report would increase the use of beta-blockers among patients with depressed left ventricular function.

Methods:

We are randomizing consecutive patients undergoing echocardiography at one of three VA echocardiography laboratories with reduced left ventricular ejection fraction (<40%) and no echocardiographic contraindication to beta-blockers (e.g. aortic stenosis) to a reminder for use of beta-blockers or to no reminder. The reminder gives starting doses for two commonly used beta-blockers (carvedilol and metoprolol). Patients are excluded from the analysis if they leave the health care system or die within three months of randomization. The primary outcome is a prescription for a beta-blocker between three and nine months following echocardiography

Status:

The project is complete.

ELIGIBILITY:
Inclusion Criteria:

Those undergoing echocardiography at one of the participating laboratories with an ejection fraction < 45%.

Exclusion Criteria:

aortic stenosis, mitral stenosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2001-05; Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Prescription for any beta-blocker

SECONDARY OUTCOMES:
Prescription for carvedilol or metoprolol succinate

CONTACTS AND LOCATIONS:
Overall Officials: Paul A. Heidenreich, MD MS, Principal Investigator — VA Palo Alto Health Care System, Palo Alto, CA
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California, United States

REFERENCES:
- [Result] Heidenreich PA, Gholami P, Sahay A, Massie B, Goldstein MK. Clinical reminders attached to echocardiography reports of patients with reduced left ventricular ejection fraction increase use of beta-blockers: a randomized trial. Circulation. 2007 Jun 5;115(22):2829-34. doi: 10.1161/CIRCULATIONAHA.106.684753. Epub 2007 May 21. PMID 17515459
- [Result] Heidenreich PA, Chacko M, Goldstein MK, Atwood JE. ACE inhibitor reminders attached to echocardiography reports of patients with reduced left ventricular ejection fraction. Am J Med. 2005 Sep;118(9):1034-7. doi: 10.1016/j.amjmed.2004.12.028. No abstract available. PMID 16164891